CLINICAL TRIAL: NCT06824246
Title: The Effect of Health Belief Model-based Water Conservation Education on Women's Water Use Behaviours: A Randomised Controlled Trial
Brief Title: The Effect of Water Conservation Education on Women's Water Use Behaviours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Deniz Kocoglu-Tanyer, Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/65
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adult Female Participants; Health Behavior; Climate Change; Water Use
Keywords: Health Belief Model; water conservation education; water footprint; water consumption habits; water consumption amount
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Parallel randomised controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: Monitoring water bill
- Intervention group (Experimental)
  Interventions: Behavioral: Water conservation education

INTERVENTIONS:
Behavioral: Water conservation education — The programme of training for participants will be based on the Health Belief Model, and will consist of two sessions on individuals' water footprints and water consumption habits. Support for the sessions will be provided by brochures and videos that have been prepared for this purpose. Women will be given brochures and a list of things to do to save water. They will also be informed that their monthly water bill will be monitored during the process.
  Arms: Intervention group
Behavioral: Monitoring water bill — Participants in the control group will be informed that their water bills will be monitored for water savings.
  Arms: Control

SUMMARY:
This research will be conducted to evaluate the effects of the Health Belief Model based water saving training prepared for women on the size of the water footprint, water consumption habits and water consumption amount. The study aims to positively change women's water consumption, water saving perceptions and beliefs, and to observe significant improvements in their knowledge levels and water consumption habits on sustainable water use.

DETAILED DESCRIPTION:
The 'water crisis' is consistently one of the top 5 global risks identified in the World Economic Forum's annual Global Risk Reports. As a result, water scarcity is rapidly becoming a global issue. The world is facing a water crisis that has reached proportions that could threaten environmental sustainability. This situation requires urgent action to protect and use water resources efficiently.

In the context of water scarcity, the promotion of awareness among individuals to minimise water usage, the modification of water consumption habits, and the enhancement of water use efficiency are of paramount importance from a public health perspective.Initiatives that predominantly advocate sustainable water conservation offer water conservation as a pivotal component of environmental initiatives. Such initiatives represent a substantial advancement for humanity in terms of planning and managing water resources in the future.The sustainable management of water is imperative for maintaining ecological balance and ensuring long-term water security. In considering the role of psychological theories in understanding and explaining human behaviour, the present research aims to examine the effect of an educational programme created using the Health Belief Model and integrated into primary care services on water use and behaviour.

The study intervention was meticulously formulated on the basis of the Health Belief Model, encompassing a training programme focused on individuals' water footprints and water consumption habits.The training programme is structured into two sessions, each spanning 30 minutes.The training programme, grounded in the Health Belief Model, encompasses the following subjects: water scarcity, water resource pollution, the ramifications of water pollution, water conservation and sustainable water utilisation. The objective of each topic is to raise awareness of water consumption, prevent water scarcity, increase compliance with water saving, reduce water consumption, and cultivate sensitivity, with the aim of effecting a change in water saving behaviours that is sustainable.The training studies were prepared by taking into account the sub-dimensions of the Health Belief Model (Sensitivity/Sensitivity Perception, Seriousness/Care Perception, Benefit Perception, Barries Perception, Actionables, Self-Efficacy).

ELIGIBILITY:
Inclusion Criteria:

* Being 20-45 years old,
* Voluntarily participating in the research,
* Household size between 3-5 people

Exclusion Criteria:

* The expectation of a rise or fall in the number of individuals residing in the dwelling at the time of the survey(due to factors such as the presence of guests or travel).

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Water consumption behavior scale | T0: The initial measurement taken prior to randomisation. T1: The final measurement taken 15 days after the conclusion of the intervention.
  The Water Consumption Behavior Scale is comprised of 16 items. The validity and reliability of the questionnaire were evaluated. The scale employs a five-point Likert type, with scores ranging from 1 to 5. The scale ranges from 16, representing the lowest attainable score, to 80, denoting the highest possible score. An increase in the score is evaluated positively.
Water footprint | T0: The initial measurement taken prior to randomisation. T1: The final measurement taken 15 days after the conclusion of the intervention.
  The water footprint, a concept developed by various non-governmental organisations and a university, is the subject of a survey comprising 14 items. It determines the amount of water individuals consume in a day (as liter) based on their water consumption habits and some nutritional habits.
Monthly water consumption amount (per person in the household) | T0: The initial measurement taken prior to randomisation. T1: The first invoice, which is issued one month after the intervention. T2: The second invoice, which is taken one month after T1.
  It will be obtained from the household's water bill.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancak Neigbourhood, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The protocol of the study will be published
Supporting Information: Study Protocol